CLINICAL TRIAL: NCT03454958
Title: Body Weight, Body Composition and Energy Balance Related Behavior During the Transition to Parenthood
Acronym: TRANSPARENTS
Status: Completed | Type: Observational
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Principal Investigator, Vicka Versele, PhD student, Vrije Universiteit Brussel
Other Study IDs: G033418N
Record Dates: First submitted 2018-02-13; First posted 2018-03-06 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Body Weight; Health Behavior; Pregnancy; First Pregnancy
MeSH Terms: conditions — Body Weight; Health Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Data collection: Data will be collected at four time points over the course of approximately one year and nine months. Participating couples (women and men) will be recruited during the first trimester of their first pregnancy. First measurement will take place in the week of the first routine ultrasound scan (week 12 of pregnancy) (=T0). First follow-up measures will take place six weeks postpartum (=T1). The second and third follow-up measurements will take place at six months postpartum (=T2) and twelve months postpartum (=T3).
  Interventions: Other: Measurements of body composition

INTERVENTIONS:
Other: Measurements of body composition — Body weight (SECA digital weighing scale), height (SECA stadiometer), body composition (TANITA Bioelectrical Impedance Analyzer & skin fold thickness measurements at the biceps, triceps, subscapular and suprailiac sites) and waist circumference (Cescorf measuring tape) will be objectively measured.

SUMMARY:
Understanding critical periods during which people are at risk to gain weight or display unhealthy changes in energy balance related behaviour, i.e. eating, physical activity and sedentary behaviour, can facilitate the development of weight gain prevention programs. Although the transition to parenthood is associated with pregnancy-related weight gain and retention in women, evidence on the effect of having a first child on men's body weight is lacking. It is also unclear whether pregnancy-related weight gain and retention cohere with unfavourable changes in body composition and energy balance related behaviour in both women and men transitioning to parenthood. Using a mixed-methods design, the investigators aim to provide insight into this critical life phase. An observational follow-up study will be used to investigate changes in body weight, body composition and energy balance related behaviour among couples from pre-conception to one year postpartum, and to identify those most at risk for excessive weight gain.

DETAILED DESCRIPTION:
The first objective of this research is to investigate both maternal and paternal changes in body weight, body composition and energy balance related behaviour during and after pregnancy in Flemish couples.

The second objective is to investigate socio-demographic and behavioural predictors of changes in both maternal and paternal body weight and body composition, in order to identify those most at risk for postpartum weight gain and retention.

Couples transitioning into parenthood (age ≥ 18 years, any BMI and socio-economic status) will be recruited during the first trimester of pregnancy by gynaecologists from the partner obstetrics units at five Flemish hospitals. All couples expecting their first child will be asked to participate in the study. Participants below 18 years of age, not speaking the Dutch language or suffering from a pathological condition that may influence energy balance related behaviour (e.g. diabetes, preeclampsia etc.) will be excluded.

Using a longitudinal design, participating couples (women and men) will be measured four times over the course of approximately one year and nine months. Baseline measurements (T0) will take place during the first trimester of pregnancy (at 12 weeks of pregnancy), with follow-up measurements at respectively six weeks (T1), and six (T2) and twelve months (T3) postpartum.

At baseline (T0), both retrospective and prospective measurements will be conducted in both pregnant women and men expecting their first child. Retrospectively, a self-report questionnaire will be used to assess body weight, height and energy balance related behaviour, incl. eating (Food Frequency Questionnaire (FFQ) which will be adapted for pregnant women), physical activity (International Physical Activity Questionnaire (IPAQ - Dutch version) and sedentary behaviour. The self-report questionnaire will also include questions about sleeping habits, smoking, and socio-demographics. Prospectively, body weight (SECA digital weighing scale), height (SECA stadiometer), body composition (TANITA Bioelectrical Impedance Analyzer & skin fold thickness measurements at the biceps, triceps, subscapular and suprailiac sites) and waist circumference (Cescorf measuring tape) will be objectively measured. Women's gestational weight will be monitored by the gynaecologists as all pregnant women are being weighed during consultation. The same self-report questionnaire (see supra) will be used prospectively, including extra questions about breastfeeding and parental leave. In addition, dietary intake will be assessed by a 3-day food diary, whereas tri-axial accelerometers (Actigraph) will be used to measure energy expenditure (by rate of physical activity and sedentary behaviour) objectively over a one-week period. At followup moments (T1-3), the same aforementioned prospective measurements will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Couples expecting their first child (nulliparous women and men)
* Participants aged ≥18 years
* Participants with any BMI
* Participants from any socio-economic status (SES)
* Participants have a sufficient proficiency of the Dutch language

Exclusion Criteria:

* Participants unable or unwilling to give informed consent
* Participants below 18 years of age
* Participants not speaking the Dutch language
* Participants suffering from a pathological condition that may influence energy balance related behaviour (e.g. diabetes,), with significant psychiatric disorder, with history of a bariatric surgery, or with requirements for complex medical diets.
* Participants who are - because of medical or other specific reasons - not allowed to exercise (e.g. bed-rest).
* Women having a multiple pregnancy (twin, triplet,…).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Couples (both men and women) will be recruited
Study Population: Couples expecting their first child
Sampling Method: Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2020-07-13 (Actual)

PRIMARY OUTCOMES:
Change in BMI | at 12 weeks of pregnancy, at 6 weeks postpartum, at 6 months postpartum, at 12 months postpartum
  Maternal and paternal body weight and height from which BMI will be calculated
Change in body composition | at 12 weeks of pregnancy, at 6 weeks postpartum, at 6 months postpartum, at 12 months postpartum
  Body composition measured by bio-electrical impedance analysis to estimate fat mass, fat free mass and muscle mass
Change in body fat | at 12 weeks of pregnancy, at 6 weeks postpartum, at 6 months postpartum, at 12 months postpartum
  Skin fold measurements for determing body fat composition by use of a skinfold calliper.
Changes in dietary intake | at 12 weeks of pregnancy, at 6 weeks postpartum, at 6 months postpartum, at 12 months postpartum
  A Food Frequency Questionnaire (FFQ) will be used for assessing dietary intake.
Change in energy expenditure | at 12 weeks of pregnancy, at 6 weeks postpartum, at 6 months postpartum, at 12 months postpartum
  Tri-axial accelerometers (Actigraph) will be used to measure energy expenditure (by ratio of physical activity and sedentary behaviour) objectively over a one-week period.
Change in physical activity | at 12 weeks of pregnancy, at 6 weeks postpartum, at 6 months postpartum, at 12 months postpartum
  Physical activity will be assessed using a self-reported questionnaire (International Physical Activity Questionnaire (IPAQ - Dutch version) and context-specific sedentary behavior.
Change in sedentary behaviour | at 12 weeks of pregnancy, at 6 weeks postpartum, at 6 months postpartum, at 12 months postpartum
  Sedentary behaviour will be assessed using a context-specific sedentary behavior questionnaire.

SECONDARY OUTCOMES:
Drop out | at 12 weeks of pregnancy, at 6 weeks postpartum, at 6 months postpartum, at 12 months postpartum
  Drop out analysis by using statistical program (SPSS)
Socio-demographics | at 12 weeks of pregnancy, at 6 weeks postpartum, at 6 months postpartum, at 12 months postpartum
  Self-reported questionnaire
Breastfeeding | at 12 weeks of pregnancy, at 6 weeks postpartum, at 6 months postpartum, at 12 months postpartum
  Self-reported questionnaire
Lifestyle behavior | at 12 weeks of pregnancy, at 6 weeks postpartum, at 6 months postpartum, at 12 months postpartum
  Self-reported questionnaire
Postnatal Depression | at 12 weeks of pregnancy, at 6 weeks postpartum, at 6 months postpartum, at 12 months postpartum
  Self-reported 23-item questionnaire
Partner support | at 12 weeks of pregnancy, at 6 weeks postpartum, at 6 months postpartum, at 12 months postpartum
  Self-reported questionnaire for social support from partner about eating and physical activity behaviour
New-borns anthropometrics | at 6 weeks postpartum, at 6 months postpartum, at 12 months postpartum
  Anthropometric measurements to determin new-borns body fat composition

CONTACTS AND LOCATIONS:
Locations (4):
- Belgium (4):
  - Ziekenhuis Oost-Limburg, Genk
  - Jessa Ziekenhuis, Hasselt
  - UZ Brussel, Jette
  - UZ Gasthuisberg, Leuven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Versele V, Stas L, Aerenhouts D, Deliens T, Matthys C, Gucciardo L, Devlieger R, Clarys P, Bogaerts A. Dietary intake, physical activity and sedentary behavior and association with BMI during the transition to parenthood: a prospective dyadic study. Front Public Health. 2023 Jun 2;11:1092843. doi: 10.3389/fpubh.2023.1092843. eCollection 2023. PMID 37333547
- [Derived] Versele V, Bogaerts A, Devlieger R, Matthys C, Gucciardo L, Deliens T, Clarys P, Aerenhouts D. Association between perceived partner support and lifestyle in mother-father dyads expecting a first child. Front Public Health. 2022 Sep 6;10:912768. doi: 10.3389/fpubh.2022.912768. eCollection 2022. PMID 36148362
- [Derived] Deliens T, Versele V, Vanden Eynde H, Clarys P, Devlieger R, Bogaerts A, Gucciardo L, Schreurs A, Van Holsbeke C, Aerenhouts D. Body weight, body composition and energy balance related behaviour during the transition to parenthood: study protocol of a multi-centre observational follow-up study (TRANSPARENTS). BMC Public Health. 2019 May 6;19(1):516. doi: 10.1186/s12889-019-6884-0. PMID 31060535